CLINICAL TRIAL: NCT04771455
Title: Testing Intervention Strategies for Addressing Obesity and Binge Eating
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Andrea Graham, Assistant Professor, Northwestern University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: STU00208056
Record Dates: First submitted 2021-02-16; First posted 2021-02-25 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Obesity; Binge Eating
MeSH Terms: conditions — Obesity; Bulimia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Condition 1 (Experimental): Behavioral weight loss intervention
  Interventions: Behavioral: Behavioral weight loss
- Condition 2 (Experimental): Behavioral weight loss intervention and decrease negative affect
  Interventions: Behavioral: Behavioral weight loss; Behavioral: Intervention component: Decrease negative affect
- Condition 3 (Experimental): Behavioral weight loss intervention and decrease unhealthy weight control practices
  Interventions: Behavioral: Behavioral weight loss; Behavioral: Intervention component: Decrease unhealthy weight control practices
- Condition 4 (Experimental): Behavioral weight loss intervention, decrease unhealthy weight control practices, and decrease negative affect
  Interventions: Behavioral: Behavioral weight loss; Behavioral: Intervention component: Decrease unhealthy weight control practices; Behavioral: Intervention component: Decrease negative affect
- Condition 5 (Experimental): Behavioral weight loss intervention and decrease overvaluation of weight and shape
  Interventions: Behavioral: Behavioral weight loss; Behavioral: Intervention component: Decrease overvaluation of weight and shape
- Condition 6 (Experimental): Behavioral weight loss intervention, decrease overvaluation of weight and shape, and decrease negative affect
  Interventions: Behavioral: Behavioral weight loss; Behavioral: Intervention component: Decrease overvaluation of weight and shape; Behavioral: Intervention component: Decrease negative affect
- Condition 7 (Experimental): Behavioral weight loss intervention, decrease overvaluation of weight and shape, and decrease unhealthy weight control practices
  Interventions: Behavioral: Behavioral weight loss; Behavioral: Intervention component: Decrease overvaluation of weight and shape; Behavioral: Intervention component: Decrease unhealthy weight control practices
- Condition 8 (Experimental): Behavioral weight loss intervention, decrease overvaluation of weight and shape, decrease unhealthy weight control practices, and decrease negative affect
  Interventions: Behavioral: Behavioral weight loss; Behavioral: Intervention component: Decrease overvaluation of weight and shape; Behavioral: Intervention component: Decrease unhealthy weight control practices; Behavioral: Intervention component: Decrease negative affect

INTERVENTIONS:
Behavioral: Behavioral weight loss — Participants will receive behavioral weight loss intervention
Behavioral: Intervention component: Decrease overvaluation of weight and shape — Participants will receive an intervention component to decrease overvaluation of weight and shape
  Arms: Condition 5; Condition 6; Condition 7; Condition 8
Behavioral: Intervention component: Decrease unhealthy weight control practices — Participants will receive an intervention component to decrease unhealthy weight control practices
  Arms: Condition 3; Condition 4; Condition 7; Condition 8
Behavioral: Intervention component: Decrease negative affect — Participants will receive an intervention component to decrease negative affect
  Arms: Condition 2; Condition 4; Condition 6; Condition 8

SUMMARY:
The purpose of this study is to conduct a randomized pilot trial of a mobile intervention that targets obesity and binge eating.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 years or older
* Obesity (BMI ≥30)
* Recurrent binge eating (≥12 episodes in the past 3 months)
* Interested in losing weight and reducing binge eating
* Willing to use a mobile application
* Has a smartphone with Internet access and capacity for calls and text messaging
* Has a valid email address
* Has access to a scale
* Not pregnant
* English-speaking

Exclusion Criteria:

* Diagnosis for which the study/intervention is not clinically indicated
* Not currently receiving clinical services for weight management or binge eating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2021-02-16 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Condition 1 | Condition 2 | Condition 3 | Condition 4 | Condition 5 | Condition 6 | Condition 7 | Condition 8
Started | 10 | 10 | 10 | 10 | 11 | 10 | 10 | 10
Completed | 9 | 9 | 8 | 9 | 11 | 8 | 10 | 9
Not Completed | 1 | 1 | 2 | 1 | 0 | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Condition 1 | Condition 2 | Condition 3 | Condition 4 | Condition 5 | Condition 6 | Condition 7 | Condition 8 | Total
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 11 | 10 | 10 | 10 | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.1 (17.6) | 36.9 (12.5) | 49.5 (10.7) | 37.5 (18.2) | 48.1 (15.3) | 41.2 (13.5) | 42.1 (15.5) | 47.3 (17.3) | 43.4 (15.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 8 | 7 | 10 | 6 | 7 | 8 | 62
  Male | 1 | 3 | 2 | 3 | 1 | 4 | 3 | 2 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 3 | 3 | 1 | 3 | 1 | 1 | 17
  Not Hispanic or Latino | 7 | 8 | 7 | 7 | 10 | 7 | 9 | 9 | 64
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Asian | 2 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 4 | 2 | 3 | 8 | 4 | 4 | 5 | 33
  White | 5 | 4 | 6 | 4 | 2 | 4 | 6 | 4 | 35
  More than one race | 0 | 0 | 1 | 3 | 0 | 1 | 0 | 0 | 5
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Weight
Description: Changes in weight
Time Frame: Measured at baseline, post-intervention (16-weeks)
Measure: Mean (Standard Deviation); unit: pounds
Groups:
- Overvaluation of Weight/Shape (Yes): Received the overvaluation of weight/shape intervention component
- Overvaluation of Weight/Shape (no): Did not receive the overvaluation of weight/shape intervention component
- Unhealthy Weight Control Practices (Yes): Received the unhealthy weight control practices intervention component
- Unhealthy Weight Control Practices (no): Did not receive the unhealthy weight control practices intervention component
- Negative Affect (Yes): Received the negative affect intervention component
- Negative Affect (no): Did not receive the negative affect intervention component
Arm/Group | Overvaluation of Weight/Shape (Yes) | Overvaluation of Weight/Shape (no) | Unhealthy Weight Control Practices (Yes) | Unhealthy Weight Control Practices (no) | Negative Affect (Yes) | Negative Affect (no)
Number analyzed (Participants) | 41 | 40 | 40 | 41 | 40 | 41
pounds | 4.2 (21.9) | 6.9 (21.3) | 4.7 (22.6) | 6.3 (20.7) | 8.5 (27.7) | 2.7 (12.6)

2. Primary Outcome: Binge Eating Episodes
Description: Changes in episodes of binge eating (past 28 days)
Time Frame: Measured at baseline, post-intervention (16-weeks)
Measure: Mean (Standard Deviation); unit: Change in number of episodes
Arm/Group | Overvaluation of Weight/Shape (Yes) | Overvaluation of Weight/Shape (no) | Unhealthy Weight Control Practices (Yes) | Unhealthy Weight Control Practices (no) | Negative Affect (Yes) | Negative Affect (no)
Number analyzed (Participants) | 41 | 40 | 40 | 41 | 40 | 41
Change in number of episodes | 8.1 (10.9) | 10.1 (13.7) | 6.9 (8.5) | 11.2 (15.0) | 9.8 (11.1) | 8.4 (13.5)

ADVERSE EVENTS:
Time Frame: 7 months
Arm/Group | Condition 1 | Condition 2 | Condition 3 | Condition 4 | Condition 5 | Condition 6 | Condition 7 | Condition 8
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10 | 0/11 | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10 | 0/11 | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10 | 0/11 | 0/10 | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-02-14): https://cdn.clinicaltrials.gov/large-docs/55/NCT04771455/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-20): https://cdn.clinicaltrials.gov/large-docs/55/NCT04771455/SAP_001.pdf